CLINICAL TRIAL: NCT05125692
Title: Vaginal Repair of Symptomatic Postcesarean Isthmocele: Evaluating A Simple Novel Technique
Brief Title: Vaginal Repair of Post Cesarean Istmocele
Acronym: OWarda
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: osama Istmocele
Record Dates: First submitted 2021-09-15; First posted 2021-11-18 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-09

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Intervention Model Description: WOMEN IN CHILDBEARING PERIOD WITH SYMPTOMATIC POSTCESAREAN ISTHMOCELE
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- women with symptomatic post cesarean Istmocele (Other): vaginal surgical repair of post cesarean symptomatic isthmocele using conventional low cost surgical techniques
  Interventions: Procedure: vaginal surgical repair of isthmocele

INTERVENTIONS:
Procedure: vaginal surgical repair of isthmocele — after preoperative identification of the borders of the isthmocele using transvaginal ultrasound measurements, the isthmocele is repaired via vaginal approach

SUMMARY:
20 WOMEN WITH SYMPTOMATIC POSTCESAREAN ISTHMOCELE (NICHE) WILL BE RECRUITED EVALUATED AND SUBJECTED TO A VAGINAL REPAIR OF THE DEFECT, RESULTS WILL BE ANALYZED.

DETAILED DESCRIPTION:
METHODS:

* Subjects: women in childbearing period with abnormal uterine bleeding or infertility attributed to post cesarean isthmocele (sample size to be calculated)
* Preoperative evaluation: transvaginal ultrasound to exclude any other uterine or adnexal pathology, and to measure:

  1. Distance from the external cervical os to the lower end of the isthmocele (A)
  2. Distance from the external cervical os to the upper end of the isthmocele(B)
  3. Length of the isthmocele (B-A)
  4. Residual myometrial thickness (the least) of the isthmocele.
* Routine preoperative workup.
* The technique:

  * Postmenstrual
  * Spinal anesthesia
  * Sterilization of the perineum and vagina
  * Cervical dilation up to 8mm using Hegar's dilators
  * Marking the previously measured points A & B
  * Making 2 transverse incisions, one 5mm below A and the other 5 mm above B.
  * The rectangular area between the 2 incisions is excised while the Hegar's dilator number 8 in in situ.
  * Hemostasis is performed using diathermy.
  * The upper and lower edges of the incision are approximated using number 2/0 vicryl on cutting needle taking 3 to 4 interrupted sutures
* The patients with uneventful postoperative course are discharged from hospital after 8 hours with doxycycline 100 mg bid for 5 days.
* Sexual intercourse is avoided for 4 weeks postoperative
* postoperative transvaginal ultrasound follow up; at 1 month postoperative.
* Data will be statistically analyzed and results will be tabulated.

ELIGIBILITY:
Inclusion Criteria:

* women diagnosed with symptomatic post cesarean isthmocele.
* should present with abnormal uterine bleeding .

Exclusion Criteria:

* presence of any other uterine pathology,
* presence of adnexal pathology,
* presence of malignancies,
* presence of pregnancy,
* presence of infection in the lower genital tract ,
* general cause of bleeding
* women not accepting the procedure,
* women not consented

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-04 (Actual); Primary Completion 2022-08-20 (Estimated); Study Completion 2022-12-20 (Estimated)

PRIMARY OUTCOMES:
myometrial thickness in supracervical area | at 1 month postoperative
  the myometrial thickness in the supracervical region is measured by transvaginal ultrasound postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospitals, Al Mansurah, Dakahlya Governorate, Egypt